CLINICAL TRIAL: NCT07288801
Title: Role of Vitamin D in Prevention of Preeclampsia Recurrence in Pregnant Women With Previous History of Preeclampsia: A Randomized Controlled Trial
Brief Title: Vitamin D for Preventing Recurrent Preeclampsia in Pregnant Women
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Dr. Tehseen Aslam, Principal Investigator, Nishtar Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U1111-1332-4347
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pre-eclampsia; Pregnancy; Vitamin D
Keywords: pre-eclampsia; pregnancy; recurrence; Vitamin D
MeSH Terms: conditions — Pre-Eclampsia; Recurrence | interventions — Vitamin D; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Oral supplementation with high dose vitamin D
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo and standard of care

INTERVENTIONS:
Drug: Vitamin D — 4000 IU of vitamin D will be given orally, once daily till 36-weeks of gestation
  Arms: Intervention
Drug: Placebo and standard of care — Look, smell and taste alike oil emulsion drops, same number, till 36-weeks of gestation
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to find out whether giving vitamin D to pregnant women who had pre-eclampsia in a previous pregnancy helps prevent the condition from coming back. The main question it aims to answer is:

Does vitamin D supplementation reduce the chance of pre-eclampsia recurring in pregnant women with a history of pre-eclampsia?

To answer this question, pregnant women attending the antenatal clinic at the Department of Obstetrics and Gynaecology, Nishtar Hospital Multan will be invited to join the study.

Participants will be randomly assigned to two equal groups:

* Vitamin D group: will take 4,000 IU of oral vitamin D until 36 weeks of gestation.
* Placebo group: will receive a pill identical in appearance, taste, and consistency but without vitamin D.

While on the study medication, each woman will visit the clinic every two weeks. At each visit, her blood pressure will be measured, and if it is 140/90 mmHg or higher, a urine test will check for protein to identify pre-eclampsia as per hospital protocol. Any diagnosis of pre-eclampsia will lead to standard care, and the outcome will be recorded.

At the end, researchers will compare how many women in each group developed recurrent pre-eclampsia.

This study will help answer whether vitamin D supplementation can safely reduce the risk of pre-eclampsia returning in women with a prior history - a question important for improving pregnancy outcomes and maternal health.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 20-weeks (on LMP method) ' - Past medical history of pre-eclampsia

Exclusion Criteria:

* Pre-existing hypertension, cardiac diseases, renal disease, thyrotoxicosis (on history and medical record)
* Women presenting with intra-uterine death of the fetus.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-08-09 (Actual); Primary Completion 2026-02-08 (Estimated); Study Completion 2026-02-08 (Estimated)

PRIMARY OUTCOMES:
Pre-eclampsia | From enrollment till 36 completed weeks of gestation
  Pregnant women, ≥ 20-weeks of gestation (on LMP method) having blood pressure of ≥140/90 mm of Hg plus protein (+1 or higher) in spot urine examination by dipstick method

CONTACTS AND LOCATIONS:
Overall Officials: Mehnaz K Professor, FCPS, Study Chair — Nishtar Medical University and Hospital
Locations (1):
- Nishtar Medical University and Hospital, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No